CLINICAL TRIAL: NCT04375592
Title: XPhe Minis - Acceptability and Tolerance Market Research
Brief Title: Acceptability and Tolerance of a Ready-to-use Protein Substitute in Tablet Form for the Dietary Management of Phenylketonuria
Status: Completed | Type: Observational
Sponsor: metaX Institut fuer Diatetik GmbH (Industry)
Collaborators: Birmingham Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XPheminisCT01
Record Dates: First submitted 2020-04-21; First posted 2020-05-05 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Phenylketonurias; Hyperphenylalaninaemia; Tetrahydrobiopterin Deficiency
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Phenylalanine-free protein substitute in tablet form (XPhe minis) — Intervention is a Phenylalanine-free protein substitute in tablet form. Subjects who currently take a concentrated second stage phenylalanine-free protein substitute will be recruited. Subjects will take the study product for 7 days and daily questionnaires will be completed. Subjects will replace some or all of their usual protein substitute with the new product. The amount of study product prescribed will be calculated to provide the same amount of protein as their usual protein substitute. Daily acceptability and tolerance questionnaires will record information on ease of preparation and administration; how it is taken; and any problems or gastrointestinal effects. Additional questions at the beginning and end of the study will record information on taste, appearance, smell, presentation and packaging of the product. Routine weekly finger prick blood spots will be collected and analysed for phenylalanine and tyrosine as usual.

SUMMARY:
The purpose of this prospective, observational study is to evaluate the tolerability and acceptability of phenylalanine-free protein substitute tablets for young children with PKU aged of 7 years or older.

DETAILED DESCRIPTION:
The principle treatment for children with phenylketonuria (PKU) is a low protein diet. Part of this treatment requires the administration of a phenylalanine-free protein substitute in order to meet basic protein requirements for normal growth and development. Several brands of phenylalanine-free protein substitutes are already available in various forms - liquid, semi solid, tablet. However, compliance with taking protein substitutes continues to be a challenge. As a low protein diet is recommended for life, long term compliance is a growing concern. As a result, improving the choice in terms of product type may aid compliance. XPhe minis are phenylalanine-free protein substitute tablets enriched with vitamins, minerals and trace elements designed for children and adults with PKU. It is anticipated that they will be a suitable alternative choice for PKU patients, broadening the variety of protein substitutes they can choose from in order to suit their lifestyle and preferences.

This is a prospective, observational tolerance study in 10 children with PKU. Subjects who are currently taking a second stage protein substitute will be recruited for a 7-day trial, taking the ready-to-use protein substitute tablets to evaluate the tolerability and acceptability of the study product. Therefore, subjects will replace some or all of their usual protein substitute with the new product.

During the 7-days trial subjects or caregivers will be asked to complete a daily questionnaire recording information on: • Usage and compliance • Ease of use and any issues with administration • Any gastro-intestinal side-effects.

A questionnaire will also be completed at the beginning and end of the study that will consider perceptions about taste, appearance, smell, ease of administration; how it is taken; and any other problems or symptoms.

The amount of tablets prescribed will be calculated to provide the same amount of protein as their usual protein substitute.

Subjects will continue to have weekly finger-prick blood tests as is routine in PKU. The results whilst on the study product will be compared with results whilst on their usual protein substitute.

10 children with PKU will be recruited. When an appropriate subject has been identified, a study information sheet will be sent to the subject or parents/caregivers. They will be invited to request further information about the study if they wish by contacting the Lead Dietitian. Recruitment of each patient will be by written informed consent, which will be completed by the parents/primary caregivers and taken by the Lead Dietitian. Children will also complete an assent/consent form and will receive an information sheet, if considered appropriate for their level of understanding.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PKU or PKU variant requiring a phenylalanine-free protein substitute.
* Subjects who are already taking a phenylalanine-free protein substitute and are willing to try the study product for 7 days.
* Children aged 7 years and over.
* Written informed consent obtained from parental caregiver.

Exclusion Criteria:

* Presence of serious concurrent illness
* Lead Dietitian's uncertainty about the willingness or ability of the patient to comply with the protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study.
* Any children having taken antibiotics over the previous 2 weeks leading up to the study.
* Children less than 7 years of age.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 10 children with PKU
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Daily compliance | 7 days
  Compliance, with currently prescribed protein substitute will be assessed at the beginning of the 7-days trial. Usage and compliance with the study product will subsequently assessed daily from days 1-7 using standardised questionnaires, where patients document the amount of consumed study product vs the prescribed doses. Compliance

SECONDARY OUTCOMES:
Treatment-Emergent tolerability | 7 days
  Gastro-intestinal side effects (including diarrhoea, constipation, bloating or abdominal distension, nausea, vomiting, burping, flatulence or regurgitation and abdominal discomfort or pain) will be assessed daily via questionnaire using the scale (none today, mild, moderate or severe / really troublesome).
Patient Acceptability | 7 days
  Acceptability (ease of use and palatability) will be assessed via questionnaire daily during the study period and at the end of the study via questionnaire .
Metabolic control | 2 days
  Weekly routine finger prick blood spots will be collected and analysed for phenylalanine (micromole per Liter) and tyrosine (micromole per Liter) as is usual clinical practice.
Incidence of study product emergent events. | Through study completion an average of 1year
  All adverse events will be recorded throughout the study (as and when they occur) and after study completion, an average of 1 year. As the study product is already commercially available occurence of any adverse event is unlikely.

CONTACTS AND LOCATIONS:
Overall Officials: Anita MacDonald, Professor, Principal Investigator — Birmingham Children´s Hospital
Locations (1):
- Birmingham Children´s Hospital, Birmingham, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual patient data will be shared with other researchers.